CLINICAL TRIAL: NCT04709575
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study Assessing the Efficacy of Anti-Bet v 1 Monoclonal Antibodies to Reduce Symptoms of Seasonal Allergic Rhinitis
Brief Title: Study to Assess the Efficacy of Anti-Bet v 1 Monoclonal Antibodies in Adults to Reduce Symptoms of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5713-5714-5715-ALG-2001; 2020-004094-52 (EudraCT Number)
Record Dates: First submitted 2020-12-23; First posted 2021-01-14 (Actual); Results first posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Allergic Rhinitis; Conjunctivitis
Keywords: Birch Allergy
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- REGN5713-5714-5715 (Experimental): REGN5713-5714-5715 administered subcutaneously
  Interventions: Drug: REGN5713; Drug: REGN5714; Drug: REGN5715
- Placebo Only (Placebo Comparator): Placebo matching REGN5713-5714-5715 administered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN5713 — Administered subcutaneously
  Arms: REGN5713-5714-5715
Drug: REGN5714 — Administered subcutaneously
  Arms: REGN5713-5714-5715
Drug: REGN5715 — Administered subcutaneously
  Arms: REGN5713-5714-5715
Drug: Placebo — Placebo that replaces REGN5713-5714-5715
  Arms: Placebo Only

SUMMARY:
The primary objective is to assess the reduction of allergic symptoms as measured by combined symptom and medication score (CSMS) during birch pollen season after a single dose of REGN5713-5714-5715 versus placebo.

ELIGIBILITY:
Key Inclusion Criteria

1. Documented or participant-reported history of birch pollen-triggered allergic rhinitis symptoms, with or without conjunctivitis, for at least 2 years
2. Positive Skin prick test (SPT) with birch pollen extract in the screening period, as defined in the protocol
3. Positive Allergen-specific IgE (sIgE) tests for birch pollen and Bet v 1 in the screening period, as defined in the protocol
4. Willing and able to comply with clinic visits and study-related procedures

Key Exclusion Criteria:

1. Participation in a prior REGN5713-5714-5715 clinical trial
2. Recurrent or chronic rhinitis or sinusitis not associated with birch pollen season, or due to daily contact with other allergens causing symptoms that are expected to coincide with birch pollen season, as assessed by the investigator
3. Participants who anticipate major changes in allergen exposure in their home or work environments that are expected to coincide with the study assessments as assessed by the investigator
4. Persistent chronic or recurring acute infection requiring treatment with antibiotics, antivirals, or antifungals, or any untreated respiratory infections (at the discretion of the investigator) within 4 weeks prior to screening visit. Participants may be re-evaluated for eligibility after symptoms resolve
5. Documentation of active SARS-CoV-2 infection, as defined in the protocol
6. A clinical history of asthma with 2 or more asthma exacerbations requiring hospitalizations or systemic corticosteroids in the previous year
7. History of birch allergy immunotherapy as defined in the protocol
8. Use of anti-IgE or other biological therapy in treatment of asthma or allergy within 6 months prior to screening

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (34):
- United States (14):
  - Regeneron Study Site, Bangor, Maine
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Plymouth, Minnesota
  - Regeneron Study Site, Columbia, Missouri
  - Regeneron Study Site, St Louis, Missouri
  - Regeneron Study Site, Missoula, Montana
  - Regeneron Study Site, Verona, New Jersey
  - Regeneron Study Site, Great Neck, New York
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Toledo, Ohio
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Pittsburgh, Pennsylvania
  - Regeneron Study Site, Lincoln, Rhode Island
  - Regeneron Study Site, Greenfield, Wisconsin
- Belgium (2):
  - Regeneron Study Site, Ghent, Oost-Vlaanderen
  - Regeneron Study Site, Leuven, Vlaams Brabant
- Canada (6):
  - Regeneron Study Site, Kingston, Ontario
  - Regeneron Study Site, London, Ontario
  - Regeneron Study Site, Ottawa, Ontario
  - Regeneron Study Site, Toronto, Ontario
  - Regeneron Study Site, Trois-Rivières, Quebec
  - Regeneron Study Site, Québec
- Denmark (3):
  - Regeneron Study Site, Hvidovre, Capital
  - Regeneron Study Site, Hellerup, Copenhagen Surroundings
  - Regeneron Study Site, Vejle, South Jutland
- Germany (9):
  - Regeneron Study Site, Heidelberg, Baden-Wurttemberg
  - Regeneron Study Site, Stuttgart, Baden-Wurttemberg
  - Regeneron Study Site, Dreieich, Hesse
  - Regeneron Study Site, Wiesbaden, Hesse
  - Regeneron Study Site, Duisburg, North Rhine-Westphalia
  - Regeneron Study Site, Düsseldorf, North Rhine-Westphalia
  - Regeneron Study Site, Dresden, Saxony
  - Regeneron Study Site, Berlin
  - Regeneron Study Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 589 participants screened, 353 randomized and from these 349 treated. 4 participants were randomized but not treated. Reasons not randomized: 235 did not meet I/E criteria, 1 withdrew consent.
Period: Overall Study
Arm/Group | REGN5713-5714-5715 | Placebo Only
Started | 176 | 177
Completed | 166 | 172
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REGN5713-5714-5715 | Placebo Only | Total
Number analyzed (Participants) | 176 | 177 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (14.15) | 42.1 (14.36) | 40.9 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 102 | 204
  Male | 74 | 75 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 172 | 174 | 346
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 10 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 165 | 161 | 326
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Combined Symptom and Medication Score (CSMS) in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Description: The average CSMS will be calculated based on daily symptom score and daily medication score recorded over the duration of the birch pollen season (BPS). CSMS is calculated by adding the Daily Medication Score (DMS) and Total Symptom Score (TSS) together, with scores ranging between 0 (none) and 38 (severe).
Time Frame: Until the end of Birch Pollen Season, up to Week 16
Population: All randomized participants with at least 1 e-diary entry with symptoms or medication score recorded during the birch pollen season.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Scores on a Scale | 7.503 (0.6545) | 8.498 (0.6534)
Statistical Analysis 1: Comparison: REGN5713-5714-5715 vs Placebo Only; Test type: Superiority; p = 0.0497, LS Mean Difference; linear mixed-effect model = -0.995, 95% CI 2-sided [-1.9886 to -0.0011]

2. Secondary Outcome: Total Symptom Score (TSS), Averaged Over the Duration of the Birch Pollen Season, in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Description: TSS is a combined score of TOSS and TNSS. TNSS and TOSS are scored as in part 1 each for a combined TSS of 0 (none) to 18 (severe)
Time Frame: Until the end of Birch Pollen Season, up to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Scores on a Scale | 5.19 (0.397) | 5.62 (0.396)

3. Secondary Outcome: Total Nasal Symptom Score (TNSS), Averaged Over the Duration of the Birch Pollen Season, in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Description: Total nasal symptom score (TNSS) is from 0 to 12 and is based on assessment of 4 nasal symptoms graded on a Likert scale ranging from 0 (none) to 3 (severe) for congestion, itching, and rhinorrhea, and from 0 (none) to 3 (5 or more sneezes) for sneezing.
Time Frame: Until the end of Birch Pollen Season, up to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Score on a scale | 3.76 (0.278) | 4.00 (0.277)

4. Secondary Outcome: Total Ocular Symptom Score (TOSS), Averaged Over the Duration of the Birch Pollen Season, in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Description: Total ocular symptom score is 0 to 6 and is based on itching/redness/gritty feeling and tearing/watering; each of the 2 symptoms is graded 0 (absent), 1 (mild), 2 (moderate), and 3 (severe)
Time Frame: Until the end of Birch Pollen Season, up to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Score on a scale | 1.43 (0.150) | 1.62 (0.150)

5. Secondary Outcome: Daily Medication Score (DMS), Averaged Over the Duration of the Birch Pollen Season, in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Description: The Daily Medication Score (DMS) is calculated by adding points for each pre-specified medication taken as follows: desloratadine 5 mg 6 points/dose; maximum daily score 6 points, olopatadine 1 mg/mL each drop 1.5 points/drop; maximum daily score 6 points, mometasone furoate 50 ug/dose 2.0 points/spray; maximum daily score 8 points). The scale is 0 (minimum) to 20 (maximum)
Time Frame: Until the end of Birch Pollen Season, up to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Score on a Scale | 2.316 (0.3993) | 2.882 (0.3986)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Throughout the Study
Description: Number of participants with any Treatment Emergent Adverse Events (TEAEs) from participating in study
Time Frame: Up to Day 127
Population: All participants in Safety Analysis Set (SAF) who received study drug and were recorded, if symptoms were displayed or not
Measure: Number; unit: Count of Participants
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 173 | 176
Count of Participants | 92 | 85

7. Secondary Outcome: Number of Participants With Serious TEAEs Throughout the Study
Description: Number of participants with any Serious Treatment Emergent Adverse Events (TEAEs) from participating in study
Time Frame: Up to Day 127
Population: as for outcome 6
Measure: Number; unit: Count of Participants
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 173 | 176
Count of Participants | 3 | 0

8. Secondary Outcome: Change From Baseline to the End of Study in Birch SPT Mean Wheal Diameter in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Description: Number of participants who showed change from baseline to the end of the study in Birch Skin Prick Test (SPT) Mean Wheal Diameter, in participants who received REGN5713-5714-5715 compared to placebo
Time Frame: Baseline through Day 127
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
millimeters | -3.139 (0.5086) | 0.553 (0.5067)

9. Secondary Outcome: Percent Change From Baseline to the End of Study in Birch SPT Mean Wheal Diameter in Participants Who Receive a Single Dose of REGN5713-5714-5715 Versus Placebo
Time Frame: Baseline through Day 127
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Percentage | -26.38 (5.179) | 8.17 (5.160)

10. Secondary Outcome: Serum Concentration of REGN5713 Over the Study Duration
Time Frame: Day 0, Day 56, Day 112
Population: All randomized and treated participants who recorded and contributed to each timepoint (+/- 14 days)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN5713-5714-5715
Number analyzed (Participants) | 172
mg/L
  Day 0 | 0 (0)
  Day 56: number analyzed (Participants) | 138
  Day 56 | 10.0 (3.97)
  Day 112: number analyzed (Participants) | 155
  Day 112 | 2.53 (1.57)

11. Secondary Outcome: Serum Concentration of REGN5714 Over the Study Duration
Time Frame: Up to Day 127
Population: All randomized and treated participants who recorded and contributed to each timepoint (+/- 14 days)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN5713-5714-5715
Number analyzed (Participants) | 172
mg/L
  Day 0 | 0 (0)
  Day 56: number analyzed (Participants) | 138
  Day 56 | 14.7 (4.68)
  Day 112: number analyzed (Participants) | 155
  Day 112 | 4.82 (2.16)

12. Secondary Outcome: Serum Concentration of REGN5715 Over the Study Duration
Time Frame: Up to Day 127
Population: All randomized and treated participants who recorded and contributed to each timepoint (+/- 14 days)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN5713-5714-5715
Number analyzed (Participants) | 172
mg/L
  Day 0 | 0 (0)
  Day 56: number analyzed (Participants) | 138
  Day 56 | 16.6 (5.34)
  Day 112: number analyzed (Participants) | 155
  Day 112 | 5.34 (2.35)

13. Secondary Outcome: Percentage of Participants With Treatment Emergent Anti-drug Antibodies to REGN5713 Throughout the Study
Description: Percentage of participants who developed antibodies to intervention provided during study
Time Frame: Up to Day 127
Population: All randomized and treated participants who recorded and contributed to each timepoint (+/- 14 days)
Measure: Number; unit: Percentage of Participants
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 168 | 171
Percentage of Participants | 0 | 0

14. Secondary Outcome: Percentage of Participants With Treatment Emergent Anti-drug Antibodies to REGN5714 Throughout the Study
Description: Percentage of participants who developed antibodies to intervention provided during study
Time Frame: Up to Day 127
Population: All randomized and treated participants who recorded and contributed to each timepoint (+/- 14 days)
Measure: Number; unit: Percentage of Participants
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 168 | 171
Percentage of Participants | 0 | 0

15. Secondary Outcome: Percentage of Participants With Treatment Emergent Anti-drug Antibodies to REGN5715 Throughout the Study
Description: Percentage of participants who developed antibodies to intervention provided during study
Time Frame: Up to Day 127
Population: All randomized and treated participants who recorded and contributed to each timepoint (+/- 14 days)
Measure: Number; unit: Percentage of Participants
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 168 | 171
Percentage of Participants | 0 | 0

16. Secondary Outcome: Number of "Well Days"
Description: "Well Days" are defined as days when rescue medication is not utilized and the Total symptom score (TSS) is ≤2/18
Time Frame: Until the end of Birch Pollen Season, up to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | REGN5713-5714-5715 | Placebo Only
Number analyzed (Participants) | 171 | 172
Days | 8.3 (1.42) | 8.6 (1.42)

ADVERSE EVENTS:
Time Frame: 28 weeks
Groups:
- Placebo: Placebo matching REGN5713-5714-5715 administered subcutaneously
- R5713-5714-5715 900 mg: REGN5713-5714-5715 administered subcutaneously
Arm/Group | Placebo | R5713-5714-5715 900 mg
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/173
Serious Adverse Events (participants affected / at risk) | 0/176 | 3/173
Other Adverse Events (participants affected / at risk) | 43/176 | 32/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=176) | R5713-5714-5715 900 mg (N=173)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=176) | R5713-5714-5715 900 mg (N=173)
Vaccination complication (Injury, poisoning and procedural complications) | 22 (29) | 17 (26)
Headache (Nervous system disorders) | 19 (22) | 15 (19)
Nasopharyngitis (Infections and infestations) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04709575/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04709575/SAP_001.pdf